CLINICAL TRIAL: NCT03106987
Title: A Phase IIIb, Randomised, Double-blind, Placebo-controlled, Multicentre Study of Olaparib Maintenance Retreatment in Patients With Epithelial Ovarian Cancer Previously Treated With a PARPi and Responding to Repeat Platinum Chemotherapy
Brief Title: A Study to Examine Olaparib Maintenance Retreatment in Patients With Epithelial Ovarian Cancer.
Acronym: OReO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D0816C00014
Record Dates: First submitted 2017-03-24; First posted 2017-04-11 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-06

CONDITIONS: Epithelial Ovarian Cancer
Keywords: polymerisation inhibitor (PARPi); PARPi re-treatment; BRCA1/2 (+ve); BRCA1/2 (-ve); Olaparib; ovarian cancer; progression free survival (PFS)
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Olaparib (Experimental): Olaparib 300mg tablets administered orally twice daily continuously.
  Interventions: Drug: Active Comparator: Olaparib tablets
- Placebo Comparator: Placebo (Placebo Comparator): Matching placebo 300mg tablets administered orally twice daily continuously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Comparator: Olaparib tablets — Olaparib
  300mg Olaparib tablets taken orally twice daily (except where this dose and formulation was previously not tolerated) until objective radiological disease progression as per RECIST 1.1 or as long as in the Investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria.
  Other Names: Olaparib tablets
  Arms: Active Comparator: Olaparib
Drug: Placebo — Placebo
  300mg placebo tablets taken orally twice daily (except where this dose and formulation was previously not tolerated) until objective radiological disease progression as per RECIST 1.1 or as long as in the Investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria.
  Arms: Placebo Comparator: Placebo

SUMMARY:
The OReO study will be a Phase IIIb, randomised, double-blind, placebo-controlled, multicentre study to assess the efficacy and tolerability of Olaparib retreatment, versus matching placebo, in non-mucinous epithelial ovarian cancer (EOC) patients (including patients with primary peritoneal and/or fallopian tube cancer)

DETAILED DESCRIPTION:
The OReO study will investigate the efficacy and safety of Olaparib maintenance re-treatment in patients with relapsed non-mucinous EOC, who have had disease progression following maintenance therapy with a Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerisation inhibitor (PARPi) and a complete or partial radiological response to subsequent treatment with platinum-based chemotherapy or may have no evidence of disease (if optimal cytoreductive surgery was conducted prior to chemotherapy), and no evidence of a rising CA-125. Patients will be enrolled on the basis of their breast cancer susceptibility gene (BRCA1, BRCA2) status into one of two cohorts (BRCA1/2 [+ve] and BRCA1/2 [-ve]). The BRCA1/2 (+ve) and BRCA1/2 (-ve) cohorts will be randomised separately. Within each cohort, patients will be randomised by prospective allocation in a 2:1 ratio (Olaparib: matching placebo).

ELIGIBILITY:
Inclusion criteria

* Provision of informed consent prior to any study specific procedures
* Female patients ≥18 years of age, with histologically diagnosed relapsed non-mucinous epithelial ovarian cancer (EOC) (including primary peritoneal and/or fallopian tube cancer) (Non-mucinous EOC includes patients with serous, endometrioid, and transitional cell tumours, and those with mixed histology where one of these subtypes is predominant (>50%). Inclusion of other subtypes should first be discussed with the Medical Monitor).
* Documented BRCA1/2 status.
* Patients must have received one prior PARPi therapy PARPi therapy includes any agent (including Olaparib) used in a maintenance setting For the BRCA1/2 (+ve) cohort, the duration of first PARPi exposure must have been ≥18 months following a first line of chemotherapy or ≥12 months following a second or subsequent line of chemotherapy For the BRCA1/2 (-ve) cohort, the duration of first PARPi exposure must have been ≥12 months following a first line of chemotherapy or ≥6 months following a second or subsequent line of chemotherapy For the last chemotherapy course immediately prior to randomisation on the study Patients must have received a platinum-based chemotherapy regimen (carboplatin, cisplatin or oxaliplatin) and have received at least 4 cycles of treatment Patients must be, in the opinion of the investigator, in response (partial or complete radiological response) or may have no evidence of disease (if optimal cytoreductive surgery was conducted prior to chemotherapy) and no evidence of a rising CA-125, as defined below, following completion of this chemotherapy course Pre-treatment CA-125 measurements must meet criterion specified below
* If the first value is within upper limit of normal (ULN) the patient is eligible to be randomised and a second sample is not required
* If the first value is greater than ULN a second assessment must be performed at least 7 days after the first. If the second assessment is ≥ 15% more than the first the patient is not eligible.

Patients must not have received bevacizumab during this course of treatment. Bevacizumab use as part of an earlier line of chemotherapy is permitted Patients must not have received any investigational agent during this course of treatment Patients must be randomised within 8 weeks of their last dose of chemotherapy (last dose is the day of the last infusion)

* Patients must have normal organ and bone marrow function measured within 28 days of randomization.
* Eastern Cooperative Oncology Group performance status 0-1
* Patients must have a life expectancy ≥16 weeks.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline with computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for repeated assessment. or No measurable disease following a complete response to most recent chemotherapy (+/- surgery)
* A formalin fixed, paraffin embedded (FFPE) tumour sample from the cancer of sufficient quantity and quality (as specified in the Covance Central Laboratory Services Manual) must be available for future central testing of tumour genetic status.
* For inclusion in the optional biomarker research, patients must sign an informed consent for biomarker research.

Exclusion criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Participation in another clinical study with an investigational product during the chemotherapy course immediately prior to randomisation.
* Other malignancy within the last 5 years except the ones detailed in the exclusion criteria section of study protocol.
* Resting electrocardiogram (ECG) with corrected QT interval (QTc) >470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome6. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative radiotherapy) within 3 weeks prior to study treatment.
* Concomitant use of known strong cytochrome P450 (CYP) subfamily 3A (CYP3A) inhibitors or moderate CYP3A inhibitors.
* Concomitant use of known strong or moderate CYP3A inducers.
* Persistent toxicities (Common Terminology Criteria for Adverse Event [CTCAE] grade 2 or higher) caused by previous cancer therapy, excluding alopecia and stable Grade 2 peripheral neuropathy .
* Patients with current or previous myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to Olaparib or any of the excipients of the product.
* Patients with a known active hepatitis (i.e..Hepatitis B or C).
* Patient who have received a whole blood transfusion within 30 days prior to screening tests (packed red blood cells and platelet transfusions are acceptable).

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pujade-Lauraine, MD, PhD, Principal Investigator — Hôpital Hôtel-Dieu
Locations (71):
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Namur
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Toronto
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, København Ø
  - Research Site, Odense C
- France (16):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (13):
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Lübeck
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Stuttgart
  - Research Site, Ulm
  - Research Site, Wiesbaden
- Israel (5):
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (10):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Candiolo
  - Research Site, Catania
  - Research Site, Lecce
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Oslo, Norway
- Poland (5):
  - Research Site, Grzepnica
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (6):
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Sutton
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Pujade-Lauraine E, Selle F, Scambia G, Asselain B, Marme F, Lindemann K, Colombo N, Madry R, Glasspool R, Vergote I, Korach J, Lheureux S, Dubot C, Oaknin A, Zamagni C, Heitz F, Gladieff L, Rubio-Perez MJ, Scollo P, Blakeley C, Shaw B, Ray-Coquard I, Redondo A; OReO/ENGOT-ov38 investigators. Maintenance olaparib rechallenge in patients with platinum-sensitive relapsed ovarian cancer previously treated with a PARP inhibitor (OReO/ENGOT-ov38): a phase IIIb trial. Ann Oncol. 2023 Dec;34(12):1152-1164. doi: 10.1016/j.annonc.2023.09.3110. Epub 2023 Oct 4. PMID 37797734
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00014&attachmentIdentifier=f6e77aa1-b549-4872-a12f-5806c419b5dd&fileName=AZ_OreO_232703_D816C00014_Final_Draft_Statistical_Analysis_Plan_to_Client_Redacted.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00014&attachmentIdentifier=59e6cde4-5803-420a-a945-6ad185f88ce7&fileName=AZ_OreO_232703_d0816c00014_Final_draft_Protocol_to_Client_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00014&attachmentIdentifier=2d40e99c-1cef-45f6-bb42-9730f35cb860&fileName=AZ_OreO_232703_d0816c00014_CSR_synopsis_Final_Draft_to_Client_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at study centres in 11 countries (France, Italy, Spain, Germany, Poland, Belgium, Denmark, Israel, United Kingdom, Norway, and Canada) between 8-Jun-2017 and 15-Feb-2021.
Pre-assignment Details: Patients were randomised into 1 of 2 cohorts depending on their known BRCA1/2 status (BRCA1/2 +ve or BRCA1/2-ve). Within each cohort, patients were randomised in a 2 Olaparib:1 placebo ratio. Randomisation was stratified by prior use of bevacizumab and number of prior regimens of platinum-containing chemotherapy.
Groups:
- Olaparib (BRCA1/2 +ve); Olaparib (BRCA1/2 -ve): Patients received olaparib 300mg tablets orally twice daily (bd) continuously
- Placebo (BRCA1/2 +ve); Placebo (BRCA1/2 -ve): Patients received placebo 300mg tablets administered orally twice daily (bd) continuously
Period: Overall Study
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Started | 74 | 38 | 72 | 36
Completed | 30 | 15 | 54 | 25
Not Completed | 44 | 23 | 18 | 11
Not completed — Death | 37 | 22 | 12 | 8
Not completed — Lost to Follow-up | 2 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 5 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomised patients analysed on an intent-to-treat (ITT) basis.
Groups:
- Placebo (BRCA +ve); Placebo (BRCA 1/2 -ve): Patients received placebo 300mg tablets administered orally twice daily (bd) continuously
- Total: Total of all reporting groups
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA 1/2 -ve) | Total
Number analyzed (Participants) | 74 | 38 | 72 | 36 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (9.31) | 61.5 (9.22) | 64.2 (9.64) | 63.3 (9.05) | 61.9 (9.54)
Age, Customized [Count of Participants; unit: Participants]
  < 50 | 11 | 3 | 4 | 1 | 19
  ≥ 50 to < 65 | 40 | 20 | 29 | 19 | 108
  ≥ 65 to < 75 | 20 | 12 | 30 | 11 | 73
  ≥ 75 | 3 | 3 | 9 | 5 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 38 | 72 | 36 | 220
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 71 | 35 | 66 | 33 | 205
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  Hawaiian Native or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 3 | 3 | 5 | 2 | 13
  Missing Data | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Progression-free Survival (PFS)
Description: PFS (per RECIST 1.1) was defined as the time from randomisation until the date of Investigator assessed objective radiological disease progression or death (by any cause in the absence of disease progression). Objective progression (per RECIST 1.1) is defined as at least a 20% increase in the sum of the diameters of the target lesions and an absolute increase of >5 mm, or an overall non-target lesion assessment of progression or a new lesion. Patients who have not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
Time Frame: At randomization visit and at every 12 weeks (+/- 7 days) until objective radiological disease progression as determined by the investigator or other discontinuation criteria are met (assessed upto 3.8 years)
Population: Full analysis set (FAS) consisted of all randomised patients analysed on an intent-to-treat (ITT) basis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Months | 4.3 [2.79 to 5.49] | 2.8 [2.73 to 4.96] | 5.3 [2.89 to 5.55] | 2.8 [2.79 to 2.89]
Statistical Analysis 1: Comparison: Olaparib (BRCA1/2 +ve) vs Placebo (BRCA1/2 +ve); Test type: Other; p = 0.0220, Stratified log-rank; Hazard Ratio (HR) = 0.566, 95% CI 2-sided [0.372 to 0.868] — Hazard Ratio (Cox Proportional Hazards model)
Statistical Analysis 2: Comparison: Olaparib (BRCA1/2 -ve) vs Placebo (BRCA1/2 -ve); Test type: Other; p = 0.0023, Stratified log-rank; Hazard Ratio (HR) = 0.430, 95% CI 2-sided [0.264 to 0.708] — Hazard Ratio (Cox Proportional Hazards model)

2. Secondary Outcome: Efficacy: Overall Survival (OS)
Description: OS was defined as the time from the date of randomisation until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive
Time Frame: From randomisation till Long-term follow-up (12-weekly beyond 30 days after last dose of study treatment) assessed upto 3.8 years
Population: FAS consisted of all randomised patients analysed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Months | 20.1 [16.39 to 25.43] | 20.9 [15.21 to 23.92] | 23.2 [15.15 to NA] — Upper limit was not calculated due to insufficient number of events. | 30.2 [17.84 to NA] — Upper limit was not calculated due to insufficient number of events.

3. Secondary Outcome: Efficacy: Time to Progression by Gynecologic Cancer Intergroup (GCIG) Criteria
Description: Time to progression by RECIST or CA-125 or death is defined as the time from randomisation to the earlier date of RECIST progression or CA-125 progression or death by any cause. Patients without a CA-125 progression or a RECIST progression who are still alive at the time of analysis will be censored at the time of their last evaluable RECIST assessment and/or their last available CA-125 measurement, whichever is the earliest at the time of analysis. Patients that do not have any evaluable RECIST assessments or any CA-125 results post-randomisation will be censored at the date of randomisation
Time Frame: At screening (Visit 1) and at every 12 weeks (±7 days), until objective disease progression, based on progressive serial elevation of serum CA-125 according to the GCIG criteria, or until discontinuation for other reasons (assessed upto 3.8 years)
Population: FAS consisted of all randomised patients analysed on an ITT basis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Months | 2.8 [2.76 to 5.36] | 2.8 [2.73 to 3.98] | 2.9 [2.79 to 5.32] | 2.79 [2.63 to 2.79]

4. Secondary Outcome: Efficacy: Time to First Subsequent Treatment Commencement (TFST)
Description: TFST was assessed as time from randomisation to first subsequent treatment commencement or death if this occurs before commencement of first subsequent treatment. Any patient not known to have had a further subsequent therapy or death was censored at the last known time to have not received subsequent therapy
Time Frame: From follow-up i.e. 30 days after last dose of study medication till end of study (assessed every 12 weeks upto 3.8 years)
Population: FAS consisted of all randomised patients analysed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Months | 5.8 [4.67 to 9.17] | 5.1 [3.58 to 6.11] | 7.9 [5.88 to 11.07] | 4.3 [3.68 to 6.41]

5. Secondary Outcome: Efficacy: Time to Second Subsequent Treatment Commencement (TSST)
Description: TSST was assessed as time from randomisation to second subsequent treatment commencement or death if this occurs before commencement of second subsequent treatment. Any patient not known to have had a further second subsequent therapy or death was censored at the last known time to have not received second subsequent therapy
Time Frame: as for outcome 4
Population: FAS consisted of all randomised patients analysed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Months | 13.1 [11.10 to 15.64] | 11.7 [8.61 to 13.60] | 15.4 [11.60 to 23.62] | 12.7 [10.35 to 16.62]

6. Secondary Outcome: Efficacy: Time to Study Treatment Discontinuation (TDT)
Description: TDT was assessed as time from randomisation to study treatment discontinuation or death if this occurs before discontinuation of study treatment. Any patient not known to have died at the time of analysis and not known to have discontinued study treatment was censored based on the last recorded date on which the patient was known to be alive
Time Frame: From follow-up 30 days after last dose of study medication till long-term follow-up i.e. 12-weekly beyond 30 days after last dose of study treatment
Population: FAS consisted of all randomised patients analysed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Months | 4.5 [3.35 to 5.59] | 3.4 [2.86 to 5.49] | 5.6 [3.42 to 5.78] | 3.1 [2.79 to 3.91]

7. Secondary Outcome: Efficacy: Change From Baseline in Health-related Quality of Life (HRQoL)
Description: Health related quality of life (HRQoL) of Olaparib maintenance retreatment compared to placebo as measured by the Functional Assessment of Cancer Therapy - Ovarian (FACT-O) Trial Outcome Index (TOI) was determined. HRQoL was analysed using the FACT-O tool by mixed model for repeated measures (MMRM) analysis of the change from baseline in TOI score. FACT-O TOI is scored from O to 100 with higher scores denoting better quality of life. The higher the score, the better the HRQoL.
Time Frame: At Baseline, and from Day 1 until objective disease progression (assessed upto 2 years)
Population: The Patient reported outcome (PRO) analysis set consisted of the FAS patients with a baseline PRO assessment
Measure: Mean (Standard Error); unit: Change in scores
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 64 | 35 | 55 | 35
Change in scores | -1.27 (0.55) | 1.67 (0.89) | -2.08 (0.60) | 0.58 (0.90)

8. Secondary Outcome: Number of Patients With Adverse Events (AEs), and Serious Adverse Events (SAEs)
Description: All AEs/serious adverse events (SAEs) reported during the study were recorded.
Time Frame: At Baseline and from Day 1 till follow-up i.e. 30 days after last dose of study medication (assessed upto 3.8 years)
Population: The safety analysis set included all patients who received at least 1 dose of randomised study treatment, Olaparib or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Participants
  Any Treatment emergent adverse event (TEAE) | 64 | 33 | 66 | 31
  Any TEAE causally related to treatment | 50 | 23 | 53 | 14
  Any TEAE of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher | 11 | 2 | 15 | 3
  Any TEAE of CTCAE grade 3 or higher, causally related to treatment | 5 | 1 | 5 | 1
  Any TEAE with outcome = death | 0 | 0 | 0 | 0
  Any TEAE with outcome = death, causally related to treatment | 0 | 0 | 0 | 0
  Any treatment-emergent SAE (including events with outcome = death) | 5 | 0 | 11 | 2
  Any treatment-emergent SAE (including events with outcome = death), causally related to treatment | 1 | 0 | 3 | 0
  Any TEAE leading to discontinuation of study medication | 2 | 0 | 1 | 0
  Any TEAE leading to discontinuation of study medication, causally related to treatment | 1 | 0 | 0 | 0
  Any TEAE leading to dose modification | 18 | 6 | 28 | 2
  Any TEAE leading to dose modification, causally related to treatment | 14 | 5 | 21 | 1

9. Secondary Outcome: Number of Patients With Adverse Event of Special Interest (AESI).
Description: All AESIs reported during the study were recorded.
Time Frame: At Baseline and from Day 1 till long-term follow-up i.e. 12-weekly beyond 30 days after last dose of study treatment (assessed upto 3.8 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
Number analyzed (Participants) | 74 | 38 | 72 | 36
Participants | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -27 to Day 0) up to 12-weekly beyond 30 days after the last dose of study treatment (assessed up to 3.8 years)
Arm/Group | Olaparib (BRCA1/2 +ve) | Placebo (BRCA1/2 +ve) | Olaparib (BRCA1/2 -ve) | Placebo (BRCA1/2 -ve)
All-Cause Mortality (participants affected / at risk) | 39/74 | 22/38 | 15/72 | 8/36
Serious Adverse Events (participants affected / at risk) | 5/74 | 0/38 | 11/72 | 2/36
Other Adverse Events (participants affected / at risk) | 64/74 | 33/38 | 65/72 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib (BRCA1/2 +ve) (N=74) | Placebo (BRCA1/2 +ve) (N=38) | Olaparib (BRCA1/2 -ve) (N=72) | Placebo (BRCA1/2 -ve) (N=36)
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Olaparib (BRCA1/2 +ve) (N=74) | Placebo (BRCA1/2 +ve) (N=38) | Olaparib (BRCA1/2 -ve) (N=72) | Placebo (BRCA1/2 -ve) (N=36)
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis cryptosporidial (Infections and infestations) | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 4 | 3 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 13 | 2 | 15 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 0 | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 0
Transplant rejection (Immune system disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 7 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0
Bell's palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 3 | 1
Dysgeusia (Nervous system disorders) | 3 | 1 | 1 | 0
Headache (Nervous system disorders) | 6 | 1 | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 2 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 4 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 2 | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 1 | 3
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 5 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 7 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 11 | 6 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 4 | 2
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0/0 | 0/0
Constipation (Gastrointestinal disorders) | 9 | 6 | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 12 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 29 | 4 | 30 | 3
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 4 | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 18 | 3 | 15 | 2
Axillary pain (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 13 | 5 | 13 | 2
Illness (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 2
Pyrexia (General disorders) | 1 | 0 | 3 | 1
Sluggishness (General disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 1 | 4 | 0
Blood urea increased (Investigations) | 2 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 0 | 3 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dyssomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cyanosis (Vascular disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 3
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03106987/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03106987/SAP_001.pdf